CLINICAL TRIAL: NCT05812976
Title: Impact of the Pulmonary Index of Microcirculatory Resistance in Pulmonary Arterial Hypertension
Brief Title: Novel Index (PIMR) in PAH
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Rushi V. Parikh, Principal Investigator, University of California, Los Angeles
Other Study IDs: IRB#22-001088
Record Dates: First submitted 2023-04-01; First posted 2023-04-14 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary Hypertension; Pulmonary Index of Microcirculatory Resistance; Pulmonary Arterial Hypertension; Index of Microcirculatory Resistance
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- PAH Patients: Pulmonary Index of Microcirculatory Resistance (PIMR) and Right Ventricle Index of Microcirculatory Resistance (RV-IMR) measurements during standard-of-care right +/- left heart catheterization at baseline and among those who undergo a standard-of-care right heart catheterization at 6 months.
  Interventions: Other: Pulmonary Index of Microcirculatory Resistance; Other: Right Ventricle Index of Microcirculatory Resistance

INTERVENTIONS:
Other: Pulmonary Index of Microcirculatory Resistance — PIMR measurement involves placing a coronary pressure wire in the pulmonary arteries and making pressure/time measurements during maximal flow down the artery.
  Other Names: PIMR
Other: Right Ventricle Index of Microcirculatory Resistance — RV-IMR measurement involves placing a coronary pressure wire in the acute marginal branch of the right coronary artery and making pressure/time measurements during maximal flow down the artery.
  Other Names: RV-IMR

SUMMARY:
The chief regulator of resistance in pulmonary arterial hypertension (PAH) is the small arteries. In the heart, the invasive measurement of the resistance of the small arteries has been shownto be safe, easy, reliable, and prognostic. This study is intended to translate prior work in heart arteries to the PAH space and invasively measure the resistance of the small arteries of the lung (pulmonary index of microcirculatory resistance [PIMR]) and the coronary artery supplying the right ventricle (acute marginal of the RCA; RV-IMR). Importantly, these measurements will be made during standard of care cardiac catheterizations (right heart catheterization [RHC] +/- left heart catheterization). The correlation between these new indices and the standard ones measured during RHC typically used to determine the severity of pulmonary hypertension will be analyzed. In addition, among newly diagnosed patients, the study will evaluate how these indices change 6 months after starting treatment. Finally, the association of these indices with clinical outcomes at 1 year will be assessed. The findings from this study may deliver an immediate impact to patient care by identifying a new metric to help better identify those who may benefit from a more intensive, personalized treatment regimen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Group 1 PAH with invasive pulmonary hypertension defined as: Mean pulmonary arterial pressure ≥ 20 mmHg, pulmonary capillary wedge pressure < 15 mmHg, and pulmonary vascular resistance ≥ 3 Wood units.
* Serum creatinine < 2.0 mg/dL
* Able to provide informed written consent

Exclusion Criteria:

* Other groups/forms of pulmonary hypertension (i.e. groups 2-5)
* Contraindicated to undergo fluoroscopy and/or coronary angiography
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult PAH patients
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
PAH hospitalization or all-cause mortality at 1 year | 1 year
  The primary outcome is the composite of PAH hospitalization or all-cause mortality at 1 year.
PIMR change from baseline | Baseline, 6 months only if repeat RHC as standard of care
  PressureWire advanced to distal third of segmental pulmonary artery (PA) for measurement of pulmonary hemodynamics. The derivation of IMR involves the application of Ohm's law (V=IR) to the coronary microcirculatory circuit, where the relationship between resistance (R) = IMR, voltage (V) = pressure (P), and current (I) = flow (Q) can be expressed as follows: IMR = ∆P/Q. ∆P = the change in pressure across the microvasculature (mean distal coronary artery pressure [Pd] - coronary venous pressure (Pv); Pv is typically disregarded because it is negligible relative to Pd. Based on the principles of thermodilution, flow is inversely proportion to mean transit time (Q ~ 1/Tmn). Lastly, the minimal achievable resistance occurs during maximal hyperemic flow when all available microvessels have theoretically been recruited. Hence, the calculation of IMR simplifies to the following formula: IMR = Pd (pulmonary artery) x TmnHyp.
RV-IMR | Baseline
  PressureWire advanced to distal third of acute marginal branch of the right coronary artery (RCA) for measurement of pulmonary hemodynamics. The derivation of IMR involves the application of Ohm's law (V=IR) to the coronary microcirculatory circuit, where the relationship between resistance (R) = IMR, voltage (V) = pressure (P), and current (I) = flow (Q) can be expressed as follows: IMR = ∆P/Q. ∆P = the change in pressure across the microvasculature (mean distal coronary artery pressure [Pd] - coronary venous pressure (Pv); Pv is typically disregarded because it is negligible relative to Pd. Based on the principles of thermodilution, flow is inversely proportion to mean transit time (Q ~ 1/Tmn). Lastly, the minimal achievable resistance occurs during maximal hyperemic flow when all available microvessels have theoretically been recruited. Hence, the calculation of IMR simplifies to the following formula: IMR = Pd (RCA marginal branch) x TmnHyp.

CONTACTS AND LOCATIONS:
Overall Officials: Rushi Parikh, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No